CLINICAL TRIAL: NCT03997461
Title: Comparison of Arterial Tonometry Sensor (BPro) With Standard Oscillometric Blood Pressure Monitoring Device (Oscar 2) for Ambulatory Use
Brief Title: Comparison of Arterial Tonometry Sensor With Standard Oscillometric Blood Pressure Monitoring Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 170706006
Record Dates: First submitted 2019-06-20; First posted 2019-06-25 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Blood Pressure
Keywords: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BPro vs Oscar 2 (Experimental): Blood pressure measurement with BPro and Oscar 2 simultaneously during 24 hours under ambulatory conditions
  Interventions: Device: BPro

INTERVENTIONS:
Device: BPro — BPro and Oscar 2 comparison for 24 hours

SUMMARY:
The study aims at comparing the values of the blood pressure measurements obtained during 24 hours by an arterial tonometry device (BPRo) and a standard oscillometric blood pressure monitoring device (Oscar 2) under ambulatory conditions

DETAILED DESCRIPTION:
The study aims at comparing the values of the blood pressure measurements obtained during 24 hours by an arterial tonometry device (BPRo) and a standard oscillometric blood pressure monitoring device (Oscar 2) under ambulatory conditions. Measurements will be taken at 15 minutes intervals during the day and 30 minutes intervals during the night.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent

Exclusion Criteria:

* Difference in blood pressure between the arms higher than 10 mmHg

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Difference in systolic blood pressure taken simultaneously by BPro and Oscar 2 devices | 24 hours
  Mean of the absolute differences in systolic blood pressure (mmHg) taken simultaneously by BPro and Oscar 2 devices at 15 minutes intervals during the day and 30 minutes intervals during the night for a period of 24 hours
Difference in diastolic blood pressure taken simultaneously by BPro and Oscar 2 devices | 24 hours
  Mean of the absolute differences in diastolic blood pressure (mmHg) taken simultaneously by BPro and Oscar 2 devices at 15 minutes intervals during the day and 30 minutes intervals during the night for a period of 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rodriguez Fernandez, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Institute for Biological and Medical Engineering, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No